CLINICAL TRIAL: NCT03443661
Title: A Pilot Phase II Study of Neoadjuvant Triplet Chemotherapy Regimen （FOLFOXIRI） in Patients With Locally Advanced Rectal Cancer
Brief Title: Neoadjuvant Triplet Chemotherapy Regimen in Patients With Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aiping Zhou (Unknown)
Responsible Party: Sponsor-Investigator, Aiping Zhou, Chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-086
Record Dates: First submitted 2018-01-14; First posted 2018-02-23 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: 5-Fluorouracil; rectal cancer; irinotecan; oxaliplatin; neoadjuvant chemotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — FOLFOXIRI protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FOLFOXIRI (Experimental): oxaliplatin 85 mg/m2 irinotecan 150 mg/m2, 5FU 2,400 mg/m2 by 46 h infusion repeated at 2week intervals
  Interventions: Drug: FOLFOXIRI

INTERVENTIONS:
Drug: FOLFOXIRI — oxaliplatin 85 mg/m2 irinotecan 150 mg/m2, 5FU 2,400 mg/m2 by 46 h infusion repeated at 2week intervals

SUMMARY:
This study aims to investigate the feasibility, safety and efficacy of triplet regimen of neoadjuvant chemotherapy in patients with locally advanced rectal cancer

DETAILED DESCRIPTION:
In this pilot phase II study, the investigators enrolled Chinese adults(age 18 to 70 years) with locally advanced stage II/III rectal cancer. The neuadjuvant chemotherapy regimen is : oxaliplatin 85 mg/m2 and irinotecan 150 mg/m2, combined with 5FU 2,400 mg/m2 by 46 h infusion, repeated at 2week intervals for 5 cycles. Total mesorectal excision was scheduled 4-5 weeks after completion of neoadjuvant treatment and followed by a further 7 cycles of mFOLFOX or 4 cycles of XELOX. Primary outcome measures of this phase II trial were feasibility, safety, tolerance and efficacy of neoadjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed locally advanced rectal cancer;
2. 18-70 years ；
3. Clinicalstage:T3,4a,N0,M0;T1-4a,N+,M0;
4. Tumor from anus >5cm and ≤15cm;
5. ECOG=0-1;
6. Available organ function:ALT≤1.5xULN;AST≤1.5xULN;TBIL≤1.0xULN; NEUT≥2×109/L;PLT≥100×109/L;Hb≥90g/L;Creatinine≤1.0xULN;
7. Informed consent;
8. UGT1A1:UGT1A1*1/UGT1A1*1,UGT1A1*1/UGT1A1*28,UGT1A1*1/UGT1A1*6;

Exclusion Criteria:

1. Clinical stage T4b or unresectable disease;
2. History of pelvic radiotherapy;
3. History of chemotherapy within 5 years;
4. History of chronic diarrhea;
5. Tumor causes intestinal obstruction, intestinal perforation, and severe bleeding;
6. Hepatitis B surface antigen positive; Hepatitis C virus infection; Cirrhosis of the liver for any cause;
7. UGT1A1:UGT1A1*28/UGT1A1*28,UGT1A1*6/UGT1A1*6;
8. Other cancers in the past 5 years, except for cervical carcinoma in situ or non-melanoma skin cancer;
9. Myocardial infarction (in the last 6 months), severe instability angina, congestive heart failure; interstitial pneumonia,pulmonary fibrosis, uncontrolled diabetes, renal insufficiency;
10. Mental illness;Pregnant or lactating women;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-02-06 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
pCR | 1 year
  Pathological complete response according to Mandard tumor regression grading

SECONDARY OUTCOMES:
R0 resection rate | 1 year
  R0 resection rate
locoregional recurrence rate | 1 year
  locoregional recurrence rate
Safety | 1 year
  Including adverse events during neoadjuvant chemotherapy,surgery and perioperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Aiping Zhou, Doctor, Principal Investigator — China National Cancer Center/Cancer Hospital, Chinese ACademy of Medical Sciences and Peking Union Medical College
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese ACademy of Medical Sciences and Peking Union Medical College, Beijing, China

REFERENCES:
- [Derived] Zhang W, Zhou H, Jiang J, Zhu Y, Zou S, Jiang L, Tang Y, Liang J, Sun Y, Jiang Z, Qu W, Li Y, Zhou A. Neoadjuvant chemotherapy with modified FOLFOXIRI for locally advanced rectal cancer to transform effectively EMVI and MRF from positive to negative: results of a long-term single center phase 2 clinical trial. BMC Cancer. 2023 Jun 27;23(1):592. doi: 10.1186/s12885-023-11103-x. PMID 37370032